CLINICAL TRIAL: NCT04910815
Title: Feasibility of a New Diagnostic Device to Assess Small Intestinal Dysbiosis in Routine Clinical Setting.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atmo Biosciences Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 72853
Record Dates: First submitted 2021-05-26; First posted 2021-06-02 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Small Intestinal Bacterial Overgrowth
MeSH Terms: interventions — Genes, fos; Breath Tests; Culture Techniques; Rifaximin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Primary recruitment (Experimental): Capsules will be ingested within 30 minutes prior to endoscopy pre- and post-antimicrobial intervention (if the patients has had a treatment) to determine if it can be used to identify increased microbial load through gas detection, and to identify responders to therapy.
  Interventions: Device: Atmo Gas Capsule; Procedure: Jejunal Aspiration and culture
- Active SIBO Arm - Rifaximin (Active Comparator): If increased microbial load is determined through culture of aspiration during initial endoscopic procedure, randomised administration of Rifaximin (550g) 1 capsule twice a day for 14 days. The post-antimicrobial endoscopic procedure will be conducted at 6 weeks post the start of treatment.
  These hydrogen concentration results will be compared to the following conventional breath tests in a crossover study design. Immediately after the endoscopic procedure, the patient will undergo a FOS challenge recording hydrogen breath samples for 2 hours in 20 min intervals while they recover from the endoscopic procedure. A standard Glucose breath test will be performed by the patients at home not earlier that 8 hours after the endoscopic procedure.
  Interventions: Device: Atmo Gas Capsule; Diagnostic Test: Glucose Breath Test; Diagnostic Test: Fructoolifosaccharides (FOS) Breath Test; Procedure: Jejunal Aspiration and culture; Drug: Rifaximin
- Active SIBO Arm - Placebo (Placebo Comparator): If increased microbial load is determined through culture of aspiration during initial endoscopic procedure, randomised administration of placebo capsule twice a day for 14 days. The placebo will be encapsulated maize starch and pregelatinised maize starch. The post-antimicrobial endoscopic procedure will be conducted at 6 weeks post the start of treatment.
  These hydrogen concentration results will be compared to the following conventional breath tests in a crossover study design. Immediately after the endoscopic procedure, the patient will undergo a FOS challenge recording hydrogen breath samples for 2 hours in 20 min intervals while they recover from the endoscopic procedure. A standard Glucose breath test will be performed by the patients at home not earlier that 8 hours after the endoscopic procedure.
  Interventions: Device: Atmo Gas Capsule; Diagnostic Test: Glucose Breath Test; Diagnostic Test: Fructoolifosaccharides (FOS) Breath Test; Procedure: Jejunal Aspiration and culture; Drug: Placebo

INTERVENTIONS:
Device: Atmo Gas Capsule — The Atmo gas capsule is an ingestible electronic device. This capsule consists of gas and temperature sensors, electronic circuits, radio transmitter and silver oxide batteries. It can measure the concentrations and types of intestinal gases in individuals and give an indication of gut transit time. This data is used for research purposes to gain an understanding of the microbiota's localised functionality. The data from the sensors is transmitted out of the body over the radio frequency to a handheld receiver. The capsule passes out of the human body at the end of the measurement and is disposable.
Diagnostic Test: Glucose Breath Test — Glucose is a sugar that will be broken down by bacteria if present in the small bowel with hydrogen gas as a by-product. The hydrogen produced through fermentation is measured in the patients exhaled breath
  Arms: Active SIBO Arm - Placebo; Active SIBO Arm - Rifaximin
Diagnostic Test: Fructoolifosaccharides (FOS) Breath Test — FOS is a long chain carbohydrate that can only be broken down by bacteria with hydrogen gas as a by-product. The hydrogen produced through fermentation is measured in the patients exhaled breath
  Arms: Active SIBO Arm - Placebo; Active SIBO Arm - Rifaximin
Procedure: Jejunal Aspiration and culture — Endoscopic procedure to determine microbial load of the Small bowel. This is the gold standard to determine the Active SIBO cases
Drug: Rifaximin — Rifaximin (550g) 1 capsule twice a day for 14 days.
  Arms: Active SIBO Arm - Rifaximin
Drug: Placebo — randomised administration of either placebo or Rifaximin (550g) 1 capsule twice a day for 14 days. The placebo will be encapsulated maize starch and pregelatinised maize starch
  Arms: Active SIBO Arm - Placebo

SUMMARY:
The purpose of this study is to determine if the gas-sensing capsule can be used to identify increased numbers and a change of the composition of microbiota or microorganisms in the gut to assess small intestinal dysbiosis

DETAILED DESCRIPTION:
In order to diagnose an increased bacterial density in the small intestine (e.g small intestinal bacterial overgrowth) metabolic activity of the microbiota colonising the small intestine is measured by exposing these bacteria with readily fermentable carbohydrates and measure subsequently (e.g. for 2 hrs) the change of the concentration of hydrogen (H2) and/or methane in the exhaled breath that results from carbohydrate fermentation in the small intestine. This is the principle of existing breath hydrogen tests, but they are poor at distinguishing where in the intestine the H2 is being produced, and their sensitivity is diminished by 'noise' in the breath H2 as a consequence of hydrogen or methane producing bacteria in the colon and this is frequently observed in the routine clinical setting. These shortcomings can be theoretically overcome by using the Atmo Gas CapsuleR which measures after ingestion gas concentrations during gastrointestinal transit in the lumen of the gut. As a consequence at the site of fermentation parts per hundred can be measured, rather than the parts per million (ppm) when methane or hydrogen are measured in the exhaled breath. An additional advantage is that the location of the capsule is known, and therefore the source of gas production from increased bacterial load can be determined. Preliminary studies using the gas capsule have shown good correlation of patterns of breath H2 with those of regional H2 patterns generated by the gas-sensing capsule. In fact, the capsule demonstrated far greater sensitivity in measuring H2 production and a vastly superior signal-to-noise ratio in response to a fermentable load than breath testing. Hence, investigating the utility of the gas-sensing capsule as a means for 'direct' assessment of microbial density presents an opportunity to overcome the shortcomings associated with the current breath test.

ELIGIBILITY:
Inclusion Criteria:

Patients aged over 18 years presenting to the Department of Gastroenterology & Hepatology at the Princess Alexandra Hospital who require and are booked for an upper gastrointestinal endoscopy as part of the routine diagnostic work up of e.g. otherwise unexplained gastrointestinal symptoms.

Exclusion Criteria:

* Radiation Enteritis
* Pregnancy
* Gastric bezoar
* Swallowing disorders/dysphagia to food or pills
* Obese, with BMI over 35
* Suspected or known strictures of the GI tract
* Fistulas or physiological/mechanical GI obstruction
* GI surgery within the past 3 months
* Diverticultis
* Patients with implantable or portable electro-mechanical medical devices, e.g. pacemakers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Structured Assessment of Gastro-Intestinal Symptoms | 30 minutes prior to endoscopy
  22 item assessing gastrointestinal symptoms. Response items are on a 5-point scale from (1 )no problem to (5) very severe problem. This is given to patients attending the Department of Gastroenterology & Hepatology at Princess Alexandra Hospital as part of their routine clinical care.
Hydrogen fermentation in the small intestine as measured by the Atmo capsule | 30 minutes prior to endoscopy
  Approximately 30 minutes before the endoscopic procedure, participants will be asked to swallow the capsule (Atmo capsule), which is the size of a large vitamin pill. If the capsule still is in the stomach at the time of the procedure it will be endoscopically pushed into the small intestine. 5g of Fructooligosaccharide (FOS) in 25mL of water will be flushed via the working channel of the endoscope into the small intestine to ensure that carbohydrates are available for fermentation. Subsequently the capsule is propelled by the normal peristaltic waves through the whole gut and is excreted after several days with the faeces. During transit the capsule transmits data about the concentration of specific gases (e.g. hydrogen) in the gut to a small receiver outside of the body.
Small Intestine microbial load as assessed by Jejunal Aspiration and Culture | During endoscpoic procedure
  The density of the bacterial colonisation of mucosal biopsies obtained during endoscpoy will be used to determine the role of the bacterial density

SECONDARY OUTCOMES:
FOS Breath samples on the day of the endoscopy | Up to 2 hours after the endescopic procedure
  Immediately prior to the endoscopy a baseline breath sample (approximately 400 cc) will be collected. FOS will be administered into the duodenum during endoscopy. After completion of the endoscopic procedure additional samples will be taken every 20 minutes up to 2 hours after the procedure.
Glucose Breath Test | Not earlier than 12 hours after the endoscopic procedure
  The patients will be asked to perform (not earlier than at least 8 hours after the endoscopic procedure) at home a standard glucose test consistent with the established clinical protocol for the diagnosis of SIBO (see SOP for Hydrogen Breath Test for Small Intestinal Bacterial Overgrowth). For this test patients will drink 75 g of glucose and breath samples will be taken at baseline and every 20 minutes for 2 hrs.
  Samples will be analysed for increased hydrogen, methane and carbon dioxide using a Breathtracker digital microlyser (Quintron Inc USA). If bacteria are present in the upper part of the small intestine, a rise in 12ppm of hydrogen over baseline is indicative of bacterial overgrowth.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Gerald Holtman, MD, PhD, MBA, Principal Investigator — The University of Queensland
Locations (2):
- Princess Alexandra Hospital, Woolloongabba, Queensland, Australia
- Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No